CLINICAL TRIAL: NCT00626028
Title: Comparison of Supplemental Oxygen and Nitric Oxide for Inhalation Plus Oxygen in the Evaluation of the Reactivity of the Pulmonary Vasculature During Acute Pulmonary Vasodilator Testing
Brief Title: Comparison of Inhaled Nitric Oxide and Oxygen in Participants Reactivity During Acute Pulmonary Vasodilator Testing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: INOT22; 2004-000625-30 (EudraCT Number)
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2016-09

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension; Cardiomyopathy
Keywords: Pulmonary Vasculature; Nitric Oxide; INOmax®; Acute Lung Injury; Pulmonary Vasodilator Testing; Idiopathic Pulmonary Arterial Hypertension; Congenital Heart Disease; reversible pulmonary hypertension; vasoreactivity; Congenital Heart Disease with Pulmonary Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Cardiomyopathies; Acute Lung Injury; Heart Defects, Congenital | interventions — Nitric Oxide; Inhalation; Endothelium-Dependent Relaxing Factors; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide First, Oxygen Last (Experimental): 10 minute dose of Nitric Oxide (NO) at 80 ppm, then 10 minute dose of NO plus Oxygen, then 10 minute washout, then 10 minute dose of 100% Oxygen on Day 1.
  Interventions: Drug: Nitric Oxide for inhalation; Drug: Oxygen; Drug: Nitric Oxide plus Oxygen
- Oxygen First, Nitric Oxide Last (Experimental): 10 minute dose of 100% Oxygen, then 10 minute dose of NO plus Oxygen, then 10 minute washout, then 10 minute dose of NO at 80 ppm on Day 1.
  Interventions: Drug: Nitric Oxide for inhalation; Drug: Oxygen; Drug: Nitric Oxide plus Oxygen

INTERVENTIONS:
Drug: Nitric Oxide for inhalation — Nitric Oxide (NO) for inhalation, given at 80ppm over 10 minutes using an INOvent® delivery system
  Other Names: INOmax®
Drug: Oxygen — 100% oxygen (O2) for inhalation, given at 80ppm over 10 minutes using an INOvent® delivery system
Drug: Nitric Oxide plus Oxygen — Nitric Oxide (NO) for inhalation plus oxygen, given at 80ppm over 10 minutes using an INOvent® delivery system
  Other Names: Inhaled Nitric Oxide, Oxygen

SUMMARY:
The primary purpose of this study is to compare the number of participants with reversible pulmonary hypertension (vasoreactivity) due to nitric oxide for inhalation and oxygen as compared to 100% oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Must have any one of these three disease categories:

   * Idiopathic Pulmonary Arterial Hypertension

     * Mean pulmonary arterial pressure (PAPm) > 25 millimeters of mercury (mmHg) at rest, pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg, and PVRI> 3 u•m^2 or diagnosed clinically with no previous catheterization
   * Congenital heart disease (CHD) with pulmonary hypertension repaired and unrepaired

     * PAPm > 25 mmHg at rest and PVRI> 3 u•m^2 or diagnosed clinically with no previous catheterization
   * Cardiomyopathy

     * PAPm > 25 mmHg at rest and Pulmonary vascular resistance index (PVRI)> 3 u•m^2 or diagnosed clinically with no previous catheterization
2. Scheduled to undergo right heart catheterization to assess pulmonary vasoreactivity by acute pulmonary vasodilation testing.
3. Male or female, ages 4 weeks to 18 years, inclusive
4. Signed informed consent/assent

Exclusion Criteria:

1. Focal pulmonary infiltrates on chest radiograph.
2. Diagnosed with severe obstructive or restrictive pulmonary disease that is significantly contributing to the patient's pulmonary hypertension.
3. Received treatment with nitric oxide for inhalation within 30 days prior to study initiation, are on other investigational medications, nitroglycerin, sodium nitroprusside, sildenafil, other Phosphodiesterase type 5 (PDE-5) inhibitors, or prostacyclin
4. Pregnant [urine human chorionic gonadotropin positive (HCG +)]
5. Baseline Pulmonary capillary wedge pressure (PCWP) > 20 mmHg

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, MD, Study Director — Mallinckrodt
Locations (18):
- United States (8):
  - Lucile Salter Packard Children's Hospital at Stanford, Stanford, California
  - The Children's Hospital, Denver, Colorado
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - New York Presbyterian Hospital, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - The Medical University of South Carolina, Charleston, South Carolina
- France (3):
  - CHU Timone - Département de cardiologie, Marseille
  - Hôpital d'Enfants, Nancy
  - Hôpital NECKER - Enfants Malades, Paris
- Beatrix Children's Hospital / University Hospital Groningen, Groningen, Netherlands
- Spain (4):
  - Hospital Sant Joan de Déu de Barcelona, Barcelona
  - Unidad de Cardiologia Infantil - Hospital Vall d'Hebrón, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Instituto Pediátrico del Corazón - Hospital Materno Infatil Doce de Octubre, Madrid
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - Southampton University Hospitals Trust - Wessex Cardiothoracic Centre, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barst RJ, Agnoletti G, Fraisse A, Baldassarre J, Wessel DL; NO Diagnostic Study Group. Vasodilator testing with nitric oxide and/or oxygen in pediatric pulmonary hypertension. Pediatr Cardiol. 2010 Jul;31(5):598-606. doi: 10.1007/s00246-010-9645-5. Epub 2010 Apr 20. PMID 20405117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children scheduled for clinically indicated right heart catheterization were screened for enrollment at 16 centers in the United States, United Kingdom, France, Spain and Netherlands.
Pre-assignment Details: All 136 patients screened received all three study drugs in a crossover design, serving as their own controls. They were randomized 1:1 into two treatment sequences.
Period: Overall Study
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Started | 68 | 68
Completed | 62 | 59
Not Completed | 6 | 9
Not completed — Adverse Event | 1 | 1
Not completed — Device Failure | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Inclusion/Exclusion Criteria | 3 | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all participants randomized regardless of actual receipt of treatment gas, the treatment gas actually received, or the appropriateness of their enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68 | 68 | 136
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (5.58) | 5.9 (5.58) | 5.9 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 34 | 34 | 68
Region of Enrollment [Number; unit: participants]
  France | 30 | 27 | 57
  United States | 15 | 17 | 32
  Spain | 12 | 12 | 24
  Netherlands | 5 | 6 | 11
  United Kingdom | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reversible Pulmonary Hypertension (Vasoreactivity)
Description: A composite of hemodynamic measurements were used to identify reversible pulmonary hypertension (vasoreactivity)
Time Frame: on Day 1
Population: All participants in the intent to treat analysis set who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Number analyzed (Participants) | 62 | 59
Participants | 28 | 16

2. Secondary Outcome: Number of Participants With Related Surgical Procedures Within 1 Year
Description: Number of participants who received surgery for pulmonary or cardiac disease within 1 year after treatment.
Time Frame: within 1 year
Population: All participants in the intent to treat analysis set who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Number analyzed (Participants) | 62 | 59
Participants | 44 | 21

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence. An AE need not have a causal relationship with treatment and included any event that was not seen at baseline or, if present at baseline, increased in severity.
Time Frame: on Day 1
Population: All participants in the intent to treat analysis set who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Number analyzed (Participants) | 62 | 59
Participants | 5 | 2

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs were collected during the 12 hours after discontinuation of gas or discharge (whichever came first). An SAE was defined as any event that resulted in death, was life threatening, resulted in permanent disability or incapacity, required or prolonged inpatient hospitalization, or was a congenital anomaly. Important medical events that, without medical or surgical intervention, would also have resulted in one of the outcomes listed above were also considered as SAEs.
Time Frame: within 12 hours
Population: Participants in the intent to treat analysis set who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Number analyzed (Participants) | 62 | 59
Participants | 3 | 0

5. Secondary Outcome: Number of Participants With Related Surgical Procedures Within 3 Years
Description: Number of participants who received surgery related to pulmonary or cardiac disease within 3 years
Time Frame: within 3 years
Population: Participants in the intent to treat population who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Number analyzed (Participants) | 62 | 59
Participants | 12 | 6

ADVERSE EVENTS:
Time Frame: within 3 years
Description: No non-serious adverse events reached the 5% reporting threshold
Arm/Group | Nitric Oxide First, Oxygen Last | Oxygen First, Nitric Oxide Last
Serious Adverse Events (participants affected / at risk) | 3/62 | 0/59
Other Adverse Events (participants affected / at risk) | 0/62 | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide First, Oxygen Last (N=62) | Oxygen First, Nitric Oxide Last (N=59)
ST Segment Elevation (Investigations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Low Cardiac Output Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Decreased oxygen saturation (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Although the first and last treatments were randomly assigned, the second treatment was always the same. Therefore, a time/treatment interaction cannot be ruled out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other